CLINICAL TRIAL: NCT00615381
Title: Clinical Trial of Euglycemia Maintenance With Supraphysiologic Insulin vs Conventional Intensive Insulin Therapy to Improve Outcomes (Neurologic, Neuropsychiatric, and Biomarkers) After Surgical Treatment of Unruptured Cerebral Aneurysms
Brief Title: Supraphysiologic Insulin to Improve Outcomes After Surgical Treatment of Unruptured Cerebral Aneurysms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not initiated and has been withdrawn due to lack of appropriate cases
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dhanesh Gupta, Associate Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DKG 2498-002
Record Dates: First submitted 2008-01-21; First posted 2008-02-14 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm, Unruptured; Craniotomy; Insulin; Neuropsychology
MeSH Terms: conditions — Intracranial Aneurysm; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal insulin (Active Comparator): Maintenance of intraoperative euglycemia (blood glucose 80--110 mg/dL) using normal intensive insulin infusion rates (0-10 U/hr).
  Interventions: Drug: Insulin
- Supraphysiologic insulin (Experimental): Maintenance of intraoperative euglycemia (blood glucose 80--110 mg/dL) using supraphysiologic insulin infusion doses (0.3 U/kg/hr) and exogenous dextrose to provide stable blood glucose levels .
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — insulin infusion (0-10 U/hr) vs. 0.3 U/kg/hr and boluses (0-8 U) adjusted every 15 minutes during the intraoperative period to maintain intraoperative euglycemia (blood glucose levels 80-120 mg/dL)
  Other Names: Novolin R (Human Recombinant Insulin)

SUMMARY:
We hypothesize that in patients undergoing surgical treatment of unruptured intracranial aneurysms, the increase in blood sugar as a result of surgical stress is detrimental to outcome, as measured by blood levels of proteins associated with systemic inflammation and 7 day, 90 day, and 1 year postoperative neurologic and neuropsychiatric outcomes. Because insulin itself is an anti-inflammatory agent, we anticipate that normalizing blood sugar levels with insulin doses higher than normally produced by the body (i.e., "supraphysiologic" insulin doses) will have a greater benefit on these outcomes than equally normalizing blood sugar levels using normal insulin doses. Based on the results of this study, we will be able to determine if a more laborious strategy to normalize blood sugar levels (i.e., "supraphysiologic" insulin therapy) offers any additional benefits to normal insulin dosing strategies. In addition, we will obtain a robust assessment of postoperative neuropsychiatric and neurologic outcomes of surgically repaired unruptured intracranial aneurysms that will serve as the basis for future studies to decrease morbidity of these patients

DETAILED DESCRIPTION:
PREOPERATIVE NEUROPSYCHIATRIC & NEUROLOGIC TESTING Up to thirty days before the scheduled elective surgical repair of his or her intracranial aneurysm, each patient will undergo neuropsychological examination by a neuropsychologist or psychometrician and assessment of neurologic status by a research nurse or the neurosurgical attending from the Department of Neurological Surgery.

The battery of neuropsychological tests will include the following:

* Benton Visual Retention Test
* Controlled Oral Word Association
* Rey-Osterrieth Complex Figure Copy
* Grooved Pegboard
* Trial Making Test
* Hopkins Verbal Learning Test

The assessment of neurologic status and the time to administer each assessment is as follows:

* Glasgow Outcome Scale (2 minutes)
* Modified Rankin Disability Scale (5 minutes)
* NIH Stroke Scale (2 minutes)

ANESTHETIC MANAGEMENT

Because of the possible effects of various anesthetic agents on immune function (in vitro and in vivo), all patients will undergo a standardized anesthetic:

1. Premedication with 0- 0.03 mg/kg midazolam
2. Induction of anesthesia with 0.05-0.5 mcg/kg/min remifentanil, 1-2 mg/kg propofol, and 0.6-1.2 mg/kg rocuronium
3. Maintenance with 0.5-0.7 MAC desflurane and 0.05-1.0 mcg/kg/min remifentanil with rocuronium 0.1-0.2 mg/kg to maintain adequate neuromuscular blockade. FIO2 = 1.0±0.1
4. Maintenance of core temperature 36.0±0.5°C
5. Propofol 50-200 mcg/kg/min to produce an EEG burst suppression ratio of 0.7-0.8 immediately before temporary occlusion of the feeding artery proximal to the intracranial aneurysm (to increase the length of time that focal ischemia is tolerated)
6. 2 mcg/kg fentanyl upon placement of the last dural stitch
7. discontinuation of desflurane and remifentanil upon removal of the head from the Mayfield head fixation
8. Postoperative analgesia with 0.2 mg dilaudid every 15 minutes, PRN
9. Antiemetic rescue with 4 mg odansetron (no standard prophylaxis)

Additional standard care & standardized therapeutics/medications are as follows:

1. Dexamethasone 10 mg after tracheal intubation followed by 4 mg every 4 hours for 48 hours
2. Mannitol 0.5-1 g/kg after completion of positioning, if requested by surgeon
3. Maintenance intravenous fluids ("4-2-1" rule) with 0.9% NaCl up to 20 mL/kg
4. Replacement of blood loss with 6% Hetastarch (1 mL : 1 mL) up to 1000 mL followed by 5% Albumin (1 mL : 1mL) up to 2500 mL
5. Nicardipine (5-15 mg/hr) ± Labetolol (5-50 mg) to keep systolic blood pressure ≤ 140 mmHg
6. Phenylephrine (10-100 mcg/min) titrated to keep systolic blood pressure ≥ 90 mmHg
7. Glycopyrollate (0.2 mg every 5 minutes) titrated to keep heart rate > 50 beats per minute

RANDOMIZATION On the day of surgery, after confirming entry into the study (i.e., confirmation of research consent and confirmation of completion of preoperative neuropsychiatric and neurologic testing), each patient will be randomly assigned to a specific protocol-Supraphysiologic Insulin vs. Normal Insulin (Appendix 1).

Randomization will be performed in blocks of 10 using a computer generated random number assignment (odd numbers = Supraphysiologic Insulin and even numbers = Normal Insulin)

MAINTENANCE OF EUGLYCEMIA Intraoperative blood glucose levels will be maintained in the target range of 80-110 mg/dL (euglycemia) using the randomly assigned protocol, as outline in Appendix 1. Blood glucose levels, insulin boluses and infusion rates, and dextrose infusion rates will be recorded on the Intraoperative Insulin & Glucose data sheet (Appendix 2).

Postoperative blood glucose levels will be maintained in the target range (80-110 mg/dL) using the standard intensive care unit protocol (Appendix 3).

PERIOPERATIVE SYSTEMIC INFLAMMATORY RESPONSE

Blood samples for serum protein analysis will be taken from the patient at the following times:

1. With the placement of the arterial line (baseline)
2. Every 4 hours after the surgical incision for 12 hours
3. 24 and 48 hours after surgical incision

When possible, the blood samples will be taken from an arterial line that is placed routinely for perioperative care. One-half (approximately 1/2) tablespoon (7 mL) of blood will be taken for plasma protein analysis at each sampling time-a total of 6 samples (approximately 3 tablespoons or 42 mL of blood) will be collected during the first 48 hours.

POSTOPERATIVE NEUROPSYCHIATRIC & NEUROLOGIC TESTING Seven days (or on discharge from the hospital) and ninety days (± 14 days) after surgery, all patients will undergo the same battery of neuropsychiatric and neurologic tests that were administered preoperatively. In addition, the SF-36 questionnaire will be administered at these times to assess the patients' sense of functional ability. Twelve months (± 30 days) after surgery, patients will be interviewed in the neurosurgeon's office or telephoned to assess neurologic recovery (using the same battery of neurologic tests administered preoperatively and the SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Unruptured intracranial aneurysm

Exclusion Criteria:

* Diabetes
* Pregnancy
* Age less than 18 years
* Inability to undergo preoperative neuropsychiatric and neurologic functional testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Neurologic Outcome--"poor" vs. "good." A "poor" outcome is assigned if the patient who arrived independently from home is discharged to a nursing home or rehabilitation hospital or dies. | Discharge from hospital after surgery

SECONDARY OUTCOMES:
Neuropsychiatric outcomes | Postoperative day 7, 90+/- 14 days, and 365+/-30 days
Neurologic Status (Glasgow Outcome Scale <=4; Modified Rankin Disability Scale >=2, NIH Stroke Scale <=10) | Postoperative day 7, 90+/- 14 days, and 365+/-30 days
Amount of time blood glucose concentration is outside the target glucose concentration range (80-120 mg/dL) | Perioperative Period (Induction of anesthesia + 24 hrs)
Biomarkers of the Perioperative Inflammatory Response | Perioperative Period (Induction of anesthesia + 48 hrs)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanesh K. Gupta, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States